CLINICAL TRIAL: NCT06379685
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of PRO-190 Ophthalmic Solution Compared to Systane Ultra® on the Ocular Surface of Ophthalmologically and Clinically Healthy Volunteers.
Brief Title: Study to Evaluate the Safety and Tolerability of PRO-190 Ophthalmic Solution Compared to Systane Ultra® on the Ocular Surface.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH190-0923/I
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye; Dry Eyes Chronic; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, comparative, controlled, comparative.
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-190 (Experimental): Propylene glycol 0.3% - Polyethylene glycol 400 0.3%. Ophthalmic solution.
  Dosage: 1 drop QID [4] (4 times per day, at least three hours apart between doses) for 7 days in both eyes,
  Route of administration: Ophthalmic.
  Interventions: Drug: PRO-190
- Systane Ultra® (Active Comparator): Propylene glycol 0.3% - Polyethylene glycol 400 0.4%. Ophthalmic solution.
  Dosage: 1 drop QID [4] (4 times per day, at least three hours apart between doses) for 7 days in both eyes,
  Route of administration: Ophthalmic.
  Interventions: Drug: Systane Ultra®

INTERVENTIONS:
Drug: PRO-190 — Propylene glycol 0.3% - Polyethylene glycol 400 0.3%. Ophthalmic solution.
  Arms: PRO-190
Drug: Systane Ultra® — Propylene glycol 0.3% - Polyethylene glycol 400 0.4%. Ophthalmic solution.
  Arms: Systane Ultra®

SUMMARY:
This is a phase I clinical study to evaluate the safety and tolerability of PRO-190 ophthalmic solution through the incidence of unexpected adverse events, changes in Best Corrected Visual Acuity (BCVA), changes in ocular surface integrity, changes in the ocular comfort index (OCI) score, and IOP measurement compared to Systane Ultra®.

DETAILED DESCRIPTION:
The variables to be evaluated include:

Primary (safety):

Incidence Unexpected Related Adverse Reactions

Secondary:

Changes in the ocular comfort index (OCI) score in between interventions Changes in Best Corrected Visual Acuity (BCVA) Changes in tear film breakup time Changes in intraocular pressure (IOP) Changes in the integrity of the ocular surface (fluorescein staining) Changes in lissamine green staining

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Clinically healthy subjects.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age ≥ 18 years.
* No history of contact lens wear
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the ied consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Having vital signs within normal parameters.
* Best corrected visual acuity (BCVA) of 20/30 or better in both eyes.
* Having an intraocular pressure ≥ 10 and ≤ 21 mmHg.

Exclusion Criteria:

* History of hypersensitivity to any of the components of the drugs under investigation.
* Use of ophthalmic medications from any pharmacological group.
* Use of medications by any other route of administration.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* History of any chronic-degenerative disease, including Diabetes Mellitus or Systemic Arterial Hypertension.
* Diagnosis of glaucoma or ocular hypertension.
* Known diagnosis of liver or heart disease.
* Presenting active inflammatory or infectious disease at the time of entry into the study.
* Presenting unresolved lesions or traumas at the time of entry into the study.
* Having been subjected to non-ophthalmological surgical procedures in the last 3 months.
* Being or having an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an employee of the research site or the sponsor, and who directly participates in this study.

Elimination Criteria

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Unexpected Related Adverse Reactions | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), 8 (Final Visit) and 12 (Safety Call) after the inclusion of each subject.
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.

SECONDARY OUTCOMES:
Changes in the ocular comfort index (OCI) score in between interventions | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  Changes in the Ocular Comfort Index (OCI) score in between interventions, the subjects will be questioned regarding this symptoms' incidence.
Changes in Best Corrected Visual Acuity (BCVA) | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  The BCVA will be evaluated through Snellen chart.
Changes in tear film breakup time | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  The most common method for assessing stability is with fluorescein. The precorneal layer colored with fluorescein will change to less fluorescent or non-fluorescent regions. The time from the last blink to the appearance of these regions is the tear film breakup time.
Changes in intraocular pressure (IOP) | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  Previous instillation of topical anesthetic, the IOP will be measured through a Goldmann tonometer during visits.
Changes in the integrity of the ocular surface (fluorescein staining) | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  Changes in the integrity of the ocular surface using fluorescein staining and evaluated through the Oxford scale. The standard Oxford scale for fluorescein staining has the following criteria: Grade 0- Equal to or less than panel A; Grade I- Equal to or less than panel B, greater than panel A; Grade II- Equal to or less than panel C, greater than panel B; Grade III- Equal or less than panel D, greater than panel C; Grade IV- Equal or less than panel E, greater than panel D; Grade V- Greater than panel E.
Changes in lissamine green staining | Through study completion, an average of 12 days. Evaluations will take place on days 0 (Basal Visit), and 8 (Final Visit) after the inclusion of each subject.
  Direct observation with slit lamp, graded according to (changes in ocular surface staining using the Sjögren's International Collaborative Clinical Alliance [SICCA].)

IPD SHARING:
Plan to Share IPD: No